CLINICAL TRIAL: NCT01719900
Title: Evaluation of Pulse Fibre Supplementation in Obesity and the Metabolic Syndrome: Generating Evidence in Support of Health Claims
Brief Title: Evaluation of Pulse Fibre Supplementation on Obesity and the Metabolic Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Alberta Innovates Health Solutions (Other); Alberta Innovates Bio Solutions (Other); Alberta Pulse Growers (Other)
Responsible Party: Principal Investigator, Dr. Raylene Reimer, Professor, Faculty of Kinesiology, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 24804
Record Dates: First submitted 2012-10-23; First posted 2012-11-01 (Estimated); Results first posted 2020-01-21 (Actual); Last update posted 2020-01-21 (Actual); Status verified 2020-01

CONDITIONS: Obesity
Keywords: Dietary intervention; Dietary fibre; Obesity; Metabolic syndrome; Weight loss; Glucose regulation; Pulse fibre
MeSH Terms: conditions — Obesity; Metabolic Syndrome; Weight Loss

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pulse Fibre (Experimental): The intervention group will receive a biscuit containing 5g/serving of yellow pea fibre to be eaten 3 times per day approximately 30 minutes prior to their 3 largest meals.
  Interventions: Dietary Supplement: Pulse fibre
- Control (Placebo Comparator): The placebo group will receive a biscuit an isocaloric control biscuit that is similar in taste and texture and without pulse fibre to be eaten 3 times per day approximately 30 minutes prior to their 3 largest meals.
  Interventions: Dietary Supplement: Control

INTERVENTIONS:
Dietary Supplement: Pulse fibre — Yellow pea hull fibre incorporated into a biscuit at 5 g/serving.
  Arms: Pulse Fibre
Dietary Supplement: Control — Control biscuit with no yellow pea hull fibre.
  Arms: Control

SUMMARY:
The recent dramatic increase in obesity has been linked to a reduction of dietary fibre intake. We hypothesized that supplementing the diet of overweight and obesity adults with pulse fibre will improve their metabolic status, chiefly defined as greater weight loss. Other metabolic health improvements may include improved glucose control and reduced inflammatory markers.

DETAILED DESCRIPTION:
The main objective of our study is to assess the effects of pulse fibre supplementation on weight loss in an overweight and obese adult population.

Primary objective - To determine the effects of a 12 week intake of 15g/day of pea hull fibre on weight loss supported by body composition measures.

Secondary objective - To measure glucose control and appetite regulation in overweight and obese adults consuming 15g/day of pea hull fibre compared to a placebo control with the use of plasma HbA1c and an oral glucose tolerance test (OGTT).

Tertiary objective - To examine mechanisms of action of pulse fibre supplementation by determining the impact of pulse fibre supplementation on gut microbiota, serum metabolomics and fecal short-chain fatty acid and bile acid concentrations.

ELIGIBILITY:
Inclusion Criteria:

* Males and females
* Age 18 - 70 years
* BMI 25 - 38 kg/m-2
* Stable body weight for at least 3 months prior to the study

Exclusion Criteria:

* Concomitant use of any weight loss medication, diet or exercise regime
* Use of corticosteroids, anti-depressants, anti-epileptic medications, lipid lowering medication, diabetes medications
* Previous bariatric or other intestinal surgeries
* Pregnancy or lactation
* Weight loss > 3 kg within preceding 3 months to enrollment
* Use of bulk laxatives or probiotics/prebiotics supplements
* Antibiotic use in the past month
* Clinically significant cardiovascular or respiratory or liver disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2012-10; Primary Completion 2013-05 (Actual); Study Completion 2018-11-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raylene Reimer, PhD, RD, Principal Investigator — University of Calgary
Locations (1):
- University of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lambert JE, Parnell JA, Han J, Sturzenegger T, Paul HA, Vogel HJ, Reimer RA. Evaluation of yellow pea fibre supplementation on weight loss and the gut microbiota: a randomized controlled trial. BMC Gastroenterol. 2014 Apr 8;14:69. doi: 10.1186/1471-230X-14-69. PMID 24712378
- [Result] Lambert JE, Parnell JA, Tunnicliffe JM, Han J, Sturzenegger T, Reimer RA. Consuming yellow pea fiber reduces voluntary energy intake and body fat in overweight/obese adults in a 12-week randomized controlled trial. Clin Nutr. 2017 Feb;36(1):126-133. doi: 10.1016/j.clnu.2015.12.016. Epub 2016 Jan 11. PMID 26811130
- [Result] Mayengbam S, Lambert JE, Parnell JA, Tunnicliffe JM, Nicolucci AC, Han J, Sturzenegger T, Shearer J, Mickiewicz B, Vogel HJ, Madsen KL, Reimer RA. Impact of dietary fiber supplementation on modulating microbiota-host-metabolic axes in obesity. J Nutr Biochem. 2019 Feb;64:228-236. doi: 10.1016/j.jnutbio.2018.11.003. Epub 2018 Nov 26. PMID 30572270

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pulse Fibre | Control
Started | 29 | 24
Completed | 22 | 22
Not Completed | 7 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pulse Fibre | Control | Total
Number analyzed (Participants) | 29 | 24 | 53
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.5 (8.1) | 44.3 (9.5) | 43.9 (14.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 20 | 43
  Male | 6 | 4 | 10
Region of Enrollment [Number; unit: participants]
  Canada | 29 | 24 | 53

OUTCOME MEASURES:

1. Primary Outcome: Change in Fat Mass at 12 Weeks
Description: Value at 12 weeks minus value at baseline assessed with dual energy x-ray absorptiometry.
Time Frame: Value at 12 weeks minus value at baseline
Measure: Mean (Standard Error); unit: kg
Arm/Group | Pulse Fibre | Control
Number analyzed (Participants) | 22 | 22
kg | -0.74 (0.26) | 0.42 (0.38)

2. Secondary Outcome: HbA1c at 12 Weeks
Description: Assessed via HbA1c
Time Frame: 12 weeks
Measure: Mean (Standard Error); unit: % in blood
Arm/Group | Pulse Fibre | Control
Number analyzed (Participants) | 22 | 22
% in blood | 5.68 (0.11) | 5.89 (0.11)

3. Secondary Outcome: Change in Objective Appetite at 12 Weeks
Description: Value at 12 weeks minus baseline energy intake during weighed lunch buffet.
Time Frame: 12 weeks minus baseline
Measure: Mean (Standard Error); unit: % of baseline food intake
Arm/Group | Pulse Fibre | Control
Number analyzed (Participants) | 22 | 22
% of baseline food intake | -16 (6) | 5 (5)

4. Other Pre Specified Outcome: Cholesterol Profile at 12 Weeks
Description: Serum LDL (low density lipoprotein) cholesterol
Time Frame: 12 weeks
Measure: Mean (Standard Error); unit: mmol/l
Arm/Group | Pulse Fibre | Control
Number analyzed (Participants) | 22 | 22
mmol/l | 2.92 (.22) | 2.90 (.21)

5. Other Pre Specified Outcome: Serum Cytokine at 12 Weeks
Description: Serum cytokine IL-6 measured at 12 weeks
Time Frame: 12 weeks
Measure: Mean (Standard Error); unit: pg/ml
Arm/Group | Pulse Fibre | Control
Number analyzed (Participants) | 22 | 22
pg/ml | 0.89 (0.20) | 1.28 (0.29)

6. Other Pre Specified Outcome: Alpha Diversity of Gut Microbiota at 12 Weeks
Description: Gut microbiota alpha diversity measured at 12 weeks as Chao index. Chao index is an abundance-based estimator of species richness within a sample. There are no preset minimum and maximum values but scores typically range from 0 to 4000. A higher score is generally regarded as better.
Time Frame: 12 weeks
Measure: Mean (Standard Error); unit: Score on a scale of 1-4000
Arm/Group | Pulse Fibre | Control
Number analyzed (Participants) | 22 | 22
Score on a scale of 1-4000 | 493 (132) | 512 (117)

7. Other Pre Specified Outcome: Serum Metabolomics at 12 Weeks
Description: Serum metabolomics measured at 12 weeks using 1H-NMR analysis. Principal component analysis is used to see if two or more groups of samples separate into distinct clusters. The principal components generated in this analysis range from 0-100%. A higher value means that more variability among the samples is explained by this principal component.
Time Frame: 12 weeks
Measure: Number; unit: score on a scale of 1-100%
Arm/Group | Pulse Fibre | Control
Number analyzed (Participants) | 22 | 22
score on a scale of 1-100% | 27 | 27

8. Other Pre Specified Outcome: Fecal Short-chain Fatty Acid Concentrations
Description: Fecal acetate concentration measured at 12 weeks
Time Frame: 12 weeks
Measure: Mean (Standard Error); unit: µmol/g dry weight
Arm/Group | Pulse Fibre | Control
Number analyzed (Participants) | 16 | 18
µmol/g dry weight | 112.7 (15.5) | 82.99 (12.97)

9. Other Pre Specified Outcome: Fecal Bile Acid Concentration
Description: Fecal cholic acid concentration measured at 12 weeks
Time Frame: 12 weeks
Measure: Mean (Standard Error); unit: µmol/g dry weight
Arm/Group | Pulse Fibre | Control
Number analyzed (Participants) | 16 | 18
µmol/g dry weight | 1.38 (0.14) | 1.99 (0.20)

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: 53 assessed for serious adverse events
Arm/Group | Pulse Fibre | Control
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/24
Other Adverse Events (participants affected / at risk) | 0/29 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No